CLINICAL TRIAL: NCT01034111
Title: An Open-label Study to Assess the Safety and Tolerability of JANUVIA (Sitagliptin) in 30 Patients With Type 2 Diabetes With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: A Local Experiential Study With Sitagliptin (an Antihyperglycemic Drug) in 30 Patients With Type 2 Diabetes Mellitus (0431-178)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431-178; 2009_705
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin (Experimental): Sitagliptin as add-on therapy to a stable dose of metformin
  Interventions: Drug: Sitagliptin phosphate; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin phosphate — Sitagliptin 100 mg tablet by mouth once daily for 4 weeks.
  Other Names: MK-0431; Januvia
Drug: Metformin — Stable dose of metformin tablet(s) by mouth (at least 1000 mg/day) for 4 weeks.
  Other Names: Glucophage

SUMMARY:
This study will assess, over a 4-week treatment period, the safety and efficacy of the addition of sitagliptin to metformin in participants with type 2 diabetes mellitus (T2DM) who failed to achieve glycemic control on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T2DM failing metformin monotherapy
* Between the ages of 18 and 79

Exclusion Criteria:

* Participants has a history of type 1 Diabetes Mellitus or ketoacidosis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-10-04 (Actual); Study Completion 2010-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitagliptin 100 mg tablet daily for 4 weeks as add-on therapy to a stable dose of metformin
Period: Overall Study
Arm/Group | Sitagliptin
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin
Number analyzed (Participants) | 30
Age, Customized [Number; unit: Participants]
  <= 40 years | 5
  41 to 50 years | 8
  51 to 60 years | 7
  >= 60 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Baseline Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 8.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Sitagliptin After 4 Weeks of Treatment
Description: Safety & tolerability were measured in terms of the # of participants with >=1 adverse event (AE), >=1 drug-related AE, >=1 serious AE (SAE), or discontinued treatment due to an AE. SAEs included events occurring after initiation of glycemic rescue therapy. AE is defined as any unfavorable/unintended change in structure, function, or chemistry of the body temporally associated with the use of SPONSOR's product. SAE is defined as any AE that results in death, is life-threatening, an overdose, causes or prolongs in-patient hospitalization, or considered medically significant by the investigator.
Time Frame: 4 weeks
Measure: Number; unit: Participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 30
Participants
  At least one adverse event | 5
  At least one drug-related adverse event | 5
  At least one serious adverse event | 0
  Discontinued treatment due to an adverse event | 0

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 4
Description: Calculated as the mean change from baseline in fasting plasma glucose at Week 4.
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin
Number analyzed (Participants) | 30
mmol/L | 1.6 (2.2)

ADVERSE EVENTS:
Arm/Group | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=30)
Hepatic Enzyme Increased (Investigations) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have the opportunity to review all abstracts, drafts or proposed presentations regarding this study 60 days prior to submission for publication/presentation. Any information that the sponsor identifies as confidential should be deleted prior to submission.